CLINICAL TRIAL: NCT02836340
Title: TIBOHCA: A Single-centre, Phase II Study to Evaluate the Safety, Tolerability and Pharmacokinetics of 2-Iminobiotin (2-IB) After Out of Hospital Cardiac Arrest
Brief Title: TIBOHCA: Safety, Tolerability and Pharmacokinetics of 2-Iminobiotin (2-IB) After OHCA
Acronym: TIBOHCA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inclusion of patients slow
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-TIBOHCA
Record Dates: First submitted 2016-06-01; First posted 2016-07-19 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Arrest; Hypoxic Ischemic Brain Injury
Keywords: neuroprotection
MeSH Terms: conditions — Heart Arrest; Hypoxia-Ischemia, Brain | interventions — 2-iminobiotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-Iminobiotin (Experimental): Increasing dosage of study drug
  Interventions: Drug: 2-Iminobiotin

INTERVENTIONS:
Drug: 2-Iminobiotin — The Investigational Medicinal Product (IMP) under study is 2-IB, which is a biotin (Vitamin H or B7) analogue and a selective inhibitor of neuronal and inducible nitric oxide synthase (NOS).

SUMMARY:
Following successful cardiopulmonary resuscitation (CPR) after out of hospital cardiac arrest (OHCA), 50% of patients admitted to the Intensive Care Unit (ICU) die. As most patients die due to brain damage sustained during cardiac arrest and the subsequent reperfusion phase, effective neuroprotective strategies could potentially improve outcome. In animal experiments, 2-Iminobiotin (2-IB), a selective neuronal and inducible nitric oxide synthase (NOS) inhibitor, given upon reperfusion has been shown to improve memory function. Since 2-IB has not shown any safety issues in preclinical and clinical studies. Before embarking on large studies with efficacy as primary endpoint, safety, tolerability and pharmacokinetics need to be established.

Objective: Evaluate short term safety and tolerability, and the pharmacokinetic properties of 2-IB in adult patients after OHCA.

Study design: Phase 2, single-centre, open-label, dose-escalation intervention study.

Study population: Three cohorts of eight evaluable patients admitted to the ICU after OHCA due to a cardiac cause.

Intervention:

The first eight patients will receive 0,055 mg/kg 2-IB every 4 hours intravenously, 6 times in total (part A). The second eight patients (cohort B) will receive 0,165 mg/kg every 4h iv, 6 times in total. The third eight patients (cohort C) will receive 0,5 mg/kg every 4h iv, 6 times in total. Medication has to be given as soon as possible and within 6h after OHCA. Escalation to the next dose level will only be done after pharmacokinetic analyses have performed, no relevant safety issues have been encountered, and the DSMB approves to move to the next dose level.

Main study parameters/endpoints:

Study parameters to evaluate short term safety and tolerability will be vital signs (heart frequency, blood pressure, cardiac ischemia) before and until 15 minutes after administration. (Serious) Adverse Events will be recorded on the ICU (up to 7 days) or until discharge from the ICU. For evaluation of the pharmacokinetics profile of 2-IB, 9 plasma samples will be analysed. Secondary parameters: Biochemical markers Neuron specific Enolase and s100b at 24h and 48h after start of study drug, occurrence of SAEs until 30 days after OHCA including death, long term term efficacy as determined by the Cerebral Performance Category (CPC), the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) or the Telephone Interview Cognitive Status (TICS) scale at 30 days after OHCA.

DETAILED DESCRIPTION:
Objective:

The primary objective of this study is to evaluate the short term safety and tolerability, and the pharmacokinetic properties of 2-IB when administered to adult patients after OHCA.

Study design:

A Phase 2, single-centre, open-label, dose-escalation intervention study.

Study population:

The study population will constitute of three cohorts of eight evaluable patients admitted to the ICU after CPR for OHCA due to a cardiac cause.

Intervention:

The first cohort of eight patients will receive 2-IB in a dose of 0,055 mg/kg/dose every 4 h iv, 6 times in total (part A). The second cohort of eight patients (cohort B) will receive an anticipated dose of 0,165 mg/kg/dose every 4h iv, 6 times in total ,and the third cohort of eight patients (cohort C) will receive an anticipated dose of 0,500 mg/kg/dose every 4h iv, 6 times in total. The first dose has to be given as soon as possible and within 6h after OHCA. Escalation to the next dose level will only be done after pharmacokinetic analyses have performed, no relevant safety issues have been encountered, and the DSMB approves to move to the next dose level.

Main study parameters/endpoints:

The main study parameters used for evaluating the short term safety and tolerability will be vital signs (heart frequency, blood pressure, cardiac ischemia) before and until 15 minutes after administration of the study drug and the need for intervention. Furthermore , biochemistry and haematology taken as part of standard clinical care will be assessed, and the occurrence of (Serious) Adverse Events ((S)AEs) until 7 days on the ICU or until discharge from the ICU, whichever occurs earlier.

For evaluation of the pharmacokinetics profile of 2-IB, 9 plasma samples will be analysed. Pharmacokinetic parameters to be determined will include Cmax, AUC, Tmax, t1/2, clearance (Cl), and volume of distribution (Vd).

Secondary parameters:

1. Short term efficacy as determined by biochemical markers NSE and s100b at 24h and 48h after start of first infusion of study drug.
2. Longer term safety as determined by the occurrence of SAEs until 30 days after OHCA including death.
3. Longer term efficacy as determined by the Cerebral Performance Category (CPC), the Computer Assisted Mild Cognitive Impairment (CAMCI) score, the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) or alternatively the Telefonisch Interview Cognitieve Status (TICS) scale (by telephone) at 30 days after OHCA.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU after OHCA and successful CPR due to a cardiac cause
* Post anoxic coma on admission
* Ability to start study medication as soon as possible, but ultimately within 6h after OHCA via a central venous line
* Age 18 years or older
* Eligible for treatment with a target temperature management of 36⁰ C

Exclusion Criteria:

* No informed consent
* Known co-morbidity with a life expectancy of <6 months prior to cardiac arrest
* Women aged 49 or less
* Severe cognitive impairment (documented dementia) known prior to OHCA
* Inability to insert a central venous line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events | 7 days
  Safety assessed as changes in heart frequency, blood pressure, cardiac ischemia (ST changes) during administration of study drug and 15 minutes thereafter and any interventions needed to maintain stability. Feasibility will be assessed by investigating whether treatment can be initiated succesfully within 6 hours after CPR.

SECONDARY OUTCOMES:
Cerebral Performance Category | 30 days
  Patients will visit the hospital or will be visited at home
Plasma levels of 2-IB | 24hours
  During the administration period nine blood samples will be taken to investigate blood levels of 2-IB
IQ-Code | 30 days
  Cognitive functioning, assessed by asking patient and caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Janneke Horn, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Intensive Care, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No